CLINICAL TRIAL: NCT05826431
Title: Feasibility, Acceptability, and Preliminary Efficacy of Cubii Under-desk Elliptical for Exercise in People With Multiple Sclerosis (PwMS)
Brief Title: Cubii for Exercise in People With MS
Acronym: Cubii
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Kevin Alschuler, Professor: Rehabilitation Medicine, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00016696
Record Dates: First submitted 2023-02-27; First posted 2023-04-24 (Actual); Results first posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Multiple Sclerosis; Fatigue; Activity, Motor; Quality of Life
MeSH Terms: conditions — Multiple Sclerosis; Fatigue; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will use the equipment for two months as they choose, keep a log of their use, and answer pre- and post- participation questionnaires.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Participants using Cubii (Experimental): Participants will use the Cubii exercise unit at their homes for two months as they choose. They will maintain a log regarding their use of the device. They will complete validated self-report questionnaires (demographics, MS disease-related variables (e.g., pain, fatigue, falls), activity, exercise, quality of life, and biopsychosocial symptom variables) before and after the use of the exercise unit.
  Interventions: Device: Cubii elliptical

INTERVENTIONS:
Device: Cubii elliptical — Low impact, portable, and compact elliptical for seated use.

SUMMARY:
The goals of this observational study are to evaluate (1) the feasibility, usability, and satisfaction with the Cubii elliptical and (2) the preliminary efficacy of the Cubii elliptical for increasing activity (primary outcome), physical function, and quality of life, and decreasing physical and psychological symptom (e.g., pain, fatigue, depression) severity in people with MS.

The main question it aims to answer is how usable and feasible is the Cubii as a mode of exercise for people with MS? Participants will use the Cubii as they choose and keep a written log of this use. They will answer questions about their demographics, MS disease-related variables (e.g., pain, fatigue, falls), activity, exercise, quality of life, and biopsychosocial symptom variables) and provide additional data regarding the feasibility, usability, and satisfaction with use of the Cubii.

DETAILED DESCRIPTION:
Data indicates people with MS are less active than their peers in the general population. Exercise interventions are important non-pharmacologic approach to maximize function and quality of life for people living with MS. Based on current evidence and expert opinion, the National Multiple Sclerosis Society (NMSS) recommends that healthcare providers promote the benefits of exercise and lifestyle physical activity for every person with MS.

Individuals with at least moderate impairments (approximately 50% of MS population) often require adaptive exercise due to mobility and balance impairments. These individuals are likely to present with neurologic impairments that impact their gait and/or coordination and may experience limitations in walking distance and necessitate precautions for falls, as well as the use of assistive devices or compensatory strategies. The Cubii product line is well-placed for this subset of the MS population because it allows for safe, seated exercise that can still meet the recommendations for aerobic and resistance training.

This study will capitalize on a representative, heterogeneous sample of MS patients who are seeking to change their coping behaviors around MS, including by exercising more, and an existing exercise unit that can be utilized by people with a range of mobility.

ELIGIBILITY:
Inclusion Criteria:

* Clinician-confirmed MS
* 18 years of age or older
* Walks with the aid of an assistive device (e.g., cane, walker, forearm crutches)
* Able to read and speak English
* Lives in the greater Seattle metropolitan area
* All genders
* Has an iPhone or Android phone that can download apps

Exclusion Criteria:

- People unable to exercise for health reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-04-19 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Alschuler, PhD, Principal Investigator — University of Washington
Locations (1):
- UW Medicine, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Participants Using Cubii
Started | 21
Completed | 20
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Participants Using Cubii
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Average Daily Use
Description: Average minutes participants used the device each day
Time Frame: Baseline - Week 9
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- Participants Using Cubii: Participants using Cubii exercise unit at their homes for two months as they choose.
Arm/Group | Participants Using Cubii
Number analyzed (Participants) | 20
Minutes | 19.72 (0.59)

2. Primary Outcome: Change in Activity - Godin Leisure Time Exercise Questionnaire
Description: The Godin Leisure-Time Exercise Questionnaire (GLTEQ; Godin & Shephard, 1985) is a 4-item self-administered questionnaire seeking information re: the number of times one engages in mild, moderate and strenuous leisure-time physical activity bouts of at least 15 min duration in a typical week. The GLTEQ was used to assess the frequency of typical weekly strenuous, moderate, and mild exercise. Total exercise scores were also computed by multiplying each reported exercise frequency by its metabolic equivalent (MET) and then summing the totals: (strenuous x 9) + (moderate x 5) + (mild x 2) (Godin, Jobin, & Boullon, 1986). Higher scores indicate greater exercise engagement.
Time Frame: [Baseline, Week 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Using Cubii
Number analyzed (Participants) | 20
units on a scale
  Baseline | 25.95 (40.73)
  Week 9 | 44.60 (85.76)
Statistical Analysis 1: Comparison: Participants Using Cubii; Study analyses were conducted using IBM SPSS Statistics Version 29. Frequencies and descriptive data were tabulated to describe the sample and quantify device use, satisfaction, and perceived impact. Qualitative responses regarding usability and feasibility were summarized based on the themes of the responses; Test type: Other; p = 0.153, Paired samples t-test; Mean Difference (Final Values) = 18.65

3. Primary Outcome: Change in Activity - Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form v2.0 - Physical Function 20a
Description: The tool asks participants to rate the difficulty in performing twenty common activities of daily living using scale that ranges from 1-5, where 1=unable to do and 5=without any difficulty.
  The total raw score is calculated by summing the individual responses. A higher score indicates higher function.
Time Frame: [Baseline, Week 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Using Cubii
Number analyzed (Participants) | 20
units on a scale
  Baseline | 40.49 (2.54)
  Week 9 | 41.10 (2.22)
Statistical Analysis 1: Comparison: Participants Using Cubii; Test type: Other; p = 0.103, Paired samples t-test; Mean Difference (Final Values) = 0.61

4. Primary Outcome: Device Utilization
Description: Qualitative findings: a narrative summary of participant responses to interview questions about using the device.
Time Frame: Baseline - Week 9
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Using Cubii
Number analyzed (Participants) | 20
Participants
  Participants reporting being very satisfied or satisfied with the Cubii as an exercise device. | 14
  Participants reporting being very likely or likely to continue to use their Cubii. | 18
  Participants reporting they were likely to recommend the device to other people with MS. | 17
  Participants reporting improvement in quality of life. | 14
  Participants reporting improvement in physical function. | 13
  Participants reporting improvement in activity level. | 14

5. Secondary Outcome: Change in Quality of Life - Multiple Sclerosis Quality of Life-54 (MSQOL54) Quality of Life Subscale
Description: A structured, self-report questionnaire examining quality of life that contains 54-items, generating 12 subscales with two summary scores (physical health and mental health) and two additional single-item measures (satisfaction with sexual function and change in health). In scoring the MSQOL-54, two summary scores (physical and mental health) are produced from a weighted combination of scale scores, where scores range from 0 to 100. A higher score indicates improved quality of life.
Time Frame: [Baseline, Week 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Using Cubii
Number analyzed (Participants) | 20
units on a scale
  Baseline | 59.74 (13.27)
  Week 9 | 63.95 (16.62)
Statistical Analysis 1: Comparison: Participants Using Cubii; Test type: Other — Single group, frequencies, and descriptive data; p = .083, Paired samples t-test; Mean Difference (Final Values) = 4.22

6. Secondary Outcome: Change in Pain Intensity - Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity Short Form 3a
Description: Patient-reported pain intensity consisting of 3 items assessing pain intensity over the past seven days. Each item is scored 1 (no pain) to 5 (very severe pain) yielding a raw score between 3 to 15, which is converted to a standard t-score. Higher scores indicate greater self-reported intensity of pain.
Time Frame: [Baseline, Week 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Using Cubii
Number analyzed (Participants) | 20
units on a scale
  Baseline | 54.21 (9.22)
  Week 9 | 53.95 (8.99)
Statistical Analysis 1: Comparison: Participants Using Cubii; Test type: Other; p = 0441, Paired samples t-test; Mean Difference (Final Values) = -0.26

7. Secondary Outcome: Change in Pain Interference - Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference Scale (Short Form 8b, V1.0)
Description: A structured, self-report questionnaire consisting of 8 items measuring the self-reported consequences of pain on relevant aspects of a person's life and may include the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities (e.g., how much did pain interfere with your day-to-day activities). Each item is scored 1 (not at all) to 5 (very much).The total raw score is calculated by summing the individual responses. The raw score ranges from 8-40; a higher score reflects more severe depressive symptoms. The total raw score is translated into a T-score for each participant according to the PROMIS Scoring Manual. The T-score provides a standardized score with a mean of 50 and a standard deviation of 10.
Time Frame: [Baseline, Week 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Using Cubii
Number analyzed (Participants) | 20
units on a scale
  Baseline | 54.72 (8.23)
  Week 9 | 57.32 (9.82)
Statistical Analysis 1: Comparison: Participants Using Cubii; Test type: Other; p = 0.095, Paired samples t-test; Mean Difference (Final Values) = 2.61

8. Secondary Outcome: Change in Fatigue Interference - Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0 - Fatigue-Multiple Sclerosis 8a
Description: A structured, self-report questionnaire consisting of 21 statements examining the effects of fatigue. Each statement is scored on a scale of 0-4 (0 = never, 1 = rarely, 2 = sometimes, 3 = often, 4 = almost always). The total MFIS score can range from 0-84; the higher the score, the stronger the feelings of fatigue.
Time Frame: [Baseline, Week 9]
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Using Cubii
Number analyzed (Participants) | 20
units on a scale
  Baseline | 59.36 (6.88)
  Week 9 | 59.39 (5.83)
Statistical Analysis 1: Comparison: Participants Using Cubii; Test type: Other; p = 0.487, Paired samples t-test; Mean Difference (Final Values) = 0.03

9. Secondary Outcome: Change in Depression - Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0 Depression 8a
Description: A structured, self-report questionnaire consisting of 8 items examining negative mood (sadness, guilt), view of self (self-criticism, worthlessness), and social cognition (loneliness, interpersonal alienation) as well as decreased positive affect and engagement (loss of interest, meaning, and purpose). Respondents rate the strength of agreement with statements about depressive symptoms using a 1-5 scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always). The total raw score is calculated by summing the individual responses. The raw score ranges from 8-40; a higher score reflects more severe depressive symptoms. The total raw score is translated into a T-score for each participant according to the PROMIS Scoring Manual. The T-score provides a standardized score with a mean of 50 and a standard deviation of 10.
Time Frame: [Baseline, Week 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Using Cubii
Number analyzed (Participants) | 20
units on a scale
  Baseline | 48.20 (11.04)
  Week 9 | 48.15 (9.51)
Statistical Analysis 1: Comparison: Participants Using Cubii; Test type: Other; p = 0.483, Paired samples t-test; Mean Difference (Final Values) = -0.06

10. Secondary Outcome: Change in Anxiety - Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form v1.0 - Anxiety 8a
Description: A structured, self-report questionnaire consisting of 6 items examining anxiety symptoms in the past 7 days using a 5-point scale (1=Never, 2=Rarely, 3=Sometimes, 4=Often, 5=Always). The lowest possible raw score is 6; the highest possible raw score is 30. Higher results mean greater anxiety symptoms. The total raw score is translated into a T-score for each participant according to the PROMIS Scoring Manual. The T-score provides a standardized score with a mean of 50 and a standard deviation of 10.
Time Frame: [Baseline, Week 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Using Cubii
Number analyzed (Participants) | 20
units on a scale
  Baseline | 48.72 (10.24)
  Week 9 | 45.90 (9.40)
Statistical Analysis 1: Comparison: Participants Using Cubii; Test type: Other; p = .0483, Paired samples t-test; Mean Difference (Final Values) = -2.82

11. Secondary Outcome: Change in Fatigue Intensity - Brief Fatigue Inventory (BFI)
Description: The BFI is a 9-item, 11-point rating scale developed to assess subjective fatigue. The first three questions measure fatigue severity from 0, indicating "no fatigue," to 10, indicating "as bad as you can imagine," at current, usual, and worst levels. The following six questions assess fatigue interference with daily activities including general activity, mood, walking ability, normal work (both inside and outside the home), relations with other people, and enjoyment of life. Response options range from 0, indicating "does not interfere," to 10, indicating, "completely interferes." Higher scores on the BFI correspond to greater self-reported levels of fatigue. The time period for all questions is over the past 24 hours.
Time Frame: [Baseline, Week 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants Using Cubii
Number analyzed (Participants) | 20
units on a scale
  Baseline | 6.60 (2.53)
  Week 9 | 6.18 (2.34)
Statistical Analysis 1: Comparison: Participants Using Cubii; Test type: Other; p = 0.123, Paired samples t-test; Mean Difference (Final Values) = -0.42

ADVERSE EVENTS:
Time Frame: 7 months and 15 days
Arm/Group | Participants Using Cubii
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
This study had limitations. As a proof-of-concept study there was no comparison group, such as a wait-list control group. While appropriate for this stage of research, the sample size was small and not generalizable. Additionally, the study timeframe was relatively short at 8 weeks; future studies would benefit from a longer follow up to assess whether use is sustained over time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-05): https://cdn.clinicaltrials.gov/large-docs/31/NCT05826431/Prot_SAP_002.pdf